CLINICAL TRIAL: NCT05001373
Title: A Phase 1, Randomized, First-in-human, Open-label Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) and Core-g28v2 60mer mRNA Vaccine (mRNA-1644v2-Core) in HIV-1 Uninfected Adults in Good General Health
Brief Title: A Phase 1 Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) and Core-g28v2 60mer mRNA Vaccine (mRNA-1644v2-Core)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: ModernaTX, Inc. (Industry); George Washington University (Other); Fred Hutchinson Cancer Center (Other); Emory University (Other); UT Health San Antonio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IAVI G002
Record Dates: First submitted 2021-07-01; First posted 2021-08-11 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Study Group 1 (Experimental): eOD-GT8 60mer mRNA Vaccine (100µg)
  Interventions: Biological: eOD-GT8 60mer mRNA Vaccine
- Study Group 2 (Experimental): eOD-GT8 60mer mRNA Vaccine (100µg) and Core-g28v2 60mer mRNA Vaccine (100µg)
  Interventions: Biological: Core-g28v2 60mer mRNA Vaccine; Biological: eOD-GT8 60mer mRNA Vaccine
- Study Group 3 (Experimental): eOD-GT8 60mer mRNA Vaccine (100µg) and Core-g28v2 60mer mRNA Vaccine (100µg)
  Interventions: Biological: Core-g28v2 60mer mRNA Vaccine; Biological: eOD-GT8 60mer mRNA Vaccine
- Study Group 4 (Experimental): Core-g28v2 60mer mRNA Vaccine (100µg)
  Interventions: Biological: Core-g28v2 60mer mRNA Vaccine

INTERVENTIONS:
Biological: Core-g28v2 60mer mRNA Vaccine — 100µg, Intramuscularly
  Arms: Study Group 2; Study Group 3; Study Group 4
Biological: eOD-GT8 60mer mRNA Vaccine — 100µg, Intramuscularly
  Arms: Study Group 1; Study Group 2; Study Group 3

SUMMARY:
A Phase 1, Randomized, First-in-human, Open-label Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) and Core-g28v2 60mer mRNA Vaccine (mRNA-1644v2-Core) in HIV-1 Uninfected Adults in Good General Health

DETAILED DESCRIPTION:
A Phase 1, Randomized, First-in-human, Open-label Study to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer mRNA Vaccine (mRNA-1644) and Core-g28v2 60mer mRNA Vaccine (mRNA-1644v2-Core) in HIV-1 Uninfected Adults in Good General Health. The hypothesis is that sequential vaccination by a germline-targeting prime followed by directional boost immunogens can induce specific classes of B-cell responses and guide their early maturation toward broadly neutralizing antibody (bnAb) development through an mRNA platform. Fifty-six participants. Adults 18 to 50 years of age who meet all protocol inclusion criteria, who do not meet any protocol exclusion criteria, who understand the study (as demonstrated by the Assessment of [Informed Consent] Understanding [AOU]), and who can provide written informed consent. Randomization allocation is 16:16:16:8 for Groups 1-4 respectively.

There is no blinding in this study. Site and study staff will not be blinded to the IP.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults as assessed by a medical history, physical examination, and laboratory tests who are at least 18 years at the time of screening and less than 51 years at the time of first IP administration;
2. Willing to comply with the requirements of the protocol and be available for follow-up for the planned duration of the study;
3. In the opinion of the Principal Investigator (PI) or designee and based on Assessment of (informed consent) Understanding (AOU) results, has understood the information provided and potential impact and/or risks linked to IP administration and participation in the study; written informed consent will be obtained from the participant before any study-related procedures are performed;
4. Willing to undergo HIV testing, risk reduction counseling, and receive HIV test results;
5. All women of reproductive potential who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception for at least 2 weeks prior to the first IP administration and continue until 4 months following the last IP administration. Effective contraception includes:

   * Condoms (male or female) with or without spermicide
   * Diaphragm or cervical cap with spermicide
   * Intrauterine device
   * Hormonal contraception, including contraceptive implant or injectable
   * Oral contraception
   * Successful vasectomy in the male partner (considered successful if a woman reports that a male partner has documentation of azoospermia by microscopy [1 year ago], or a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy)
   * Not of reproductive potential, such as having undergone hysterectomy, bilateral oophorectomy or tubal ligation, postmenopausal (≥45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/L), surgically sterile Note: More restrictive measures may be required by the study sites.
6. All participants born female who are not heterosexually active at screening must agree to utilize an effective method of contraception if they become heterosexually active as outlined above;
7. All participants born female who are of reproductive potential must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Activities (SOA);
8. All sexually active participants born male, regardless of reproductive potential, must be willing to use an effective method of contraception (such as consistent condom use) from the day of the first IP administration until at least 4 months after the last IP administration;
9. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to IP-induced antibodies, until the anti-HIV antibody titers become undetectable.

Exclusion Criteria:

1. Positive test for HIV-1 or HIV-2;
2. Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, antituberculosis, or other medications considered significant by the Investigator within the previous 6 months; Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis, or a short course (duration of 10 days or less or a single injection) of corticosteroid for a non-chronic condition (based on Investigator's clinical judgment) at least 2 weeks prior to enrolment in this study.
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the Investigator makes the participant unsuitable for participation in the study; Note: All chronic conditions must be considered stable, there can be no significant change of medications within the previous 2 months, and for diabetics HgbA1c must be <10%.
4. History of substance abuse or alcohol abuse;
5. Reported behavior that puts the participant at risk for HIV infection within 6 months prior to screening, as defined by:

   * Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection, or a casual partner (ie, no continuing established relationship)
   * Engaged in sex work
   * Frequent excessive daily alcohol use or frequent binge drinking, or any other use of illicit drugs
   * History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus-2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B-or hepatitis C;
   * Three or more sexual partners
6. If female, pregnant or planning a pregnancy during the period of enrolment until 4 months after the last IP administration; or lactating;
7. Bleeding disorder that was diagnosed by a physician (eg, factor deficiency, coagulopathy, or platelet disorder that requires special precautions) Note: A participant who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has IM vaccinations and blood draws without any adverse experience is eligible;
8. Infectious disease diagnosis: chronic hepatitis B-infection (HBsAg-positive), current hepatitis C infection (HCV Ab-positive and HCV RNA positive), or active syphilis (screening and confirmatory tests);
9. History of splenectomy;
10. Any of the following abnormal laboratory parameters listed below at screening:

    Hematology
    * Hemoglobin ≤10.5 g/dl or ≤6.5 mmol/L in females; ≤11.0 g/dl or ≤6.8 mmol/L in males
    * Absolute Neutrophil Count (ANC) ≤1,000/mm3 or ≤1.0 × 109 cells/L
    * Absolute Lymphocyte Count (ALC) ≤650/mm3 or ≤0.65 × 109 cells/L
    * Platelets ≤125,000 cells/mm3 or ≤125 × 109 cells/L Chemistry
    * Creatinine ≥1.1 × upper limit of normal (ULN)
    * AST ≥1.25 × ULN
    * ALT ≥1.25 × ULN Urinalysis

    Clinically significant abnormal dipstick confirmed by microscopy:

    • Protein = 1 + or more Blood = 2 + or more (not due to menses) or >10 RBCs per high power field. If Urinalysis is the only exclusion criteria that is met, consider repeat urinalysis to confirm
11. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after IP administration; or receipt of other vaccine (including all authorized or approved COVID-19 vaccinations) within the previous 14 days or planned receipt within 14 days after IP administration. (Exception is live attenuated influenza vaccine within 14 days); Note 1: COVID-19 vaccinations: Participants should not have received any COVID-19 vaccinations in the 14 days before or 14 days after IP administration.

    Note 2: COVID-19 immunoprophylaxis will be permitted prior to and/or during the study provided the agent has received either Emergency Use Approval from FDA, Conditional Marketing Authorization from EMA, or granted licensure from a country's regulatory agency.
12. Receipt of blood transfusion or blood-derived products within the previous 3 months;
13. Participation in another clinical study of an IP currently, within the previous 3 months or expected participation during this study; Note: Concurrent participation in an observational study not requiring blood or tissue sample collection is not an exclusion;
14. Prior receipt of any investigational HIV vaccine candidate or HIV monoclonal antibody; Note: Receipt of placebo in a previous monoclonal antibody including HIV monoclonal antibody study will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval.
15. History of significant local or systemic reactogenicity to vaccines (eg, anaphylaxis, respiratory difficulties, angioedema, injection site necrosis, or ulceration); (This includes individuals with history of anaphylaxis and/or severe hypersensitivity reaction to mRNA vaccines or its excipients)
16. Psychiatric condition that compromises the safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years;
17. Seizure disorder: A participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years);
18. History of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of completely excised malignancy that is considered cured is not an exclusion);
19. Active, serious infections as assessed by the Investigator requiring antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment;
20. Body mass index (BMI) ≥35;
21. Body weight <110 pounds (50 kg);
22. Prior daily use of NSAID/aspirin that cannot be held for 5 days prior to the leukapheresis procedure (if applicable at the study site);
23. If, in the opinion of the PI, it is not in the best interest of the participant to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 9 months
  * Proportion of participants with local and systemic solicited Adverse Events (AEs) from Day 1 to Day 7 inclusive after each IP administration
  * Proportion of participants with Grade 2 or higher unsolicited Adverse Events (AEs), including safety laboratory (biochemical, hematological) parameters from the day of each IP administration through 28 days after each IP administration (any event AND any possibly, probably, or definitely related event)
  * Proportion of participants with Serious Adverse Events (SAEs) throughout the study period (any event AND any possibly, probably, or definitely related event)
  * Proportion of participants with Medical Attended Adverse Events (MAAEs) from the first day of IP administration through 24 weeks post final IP administration

SECONDARY OUTCOMES:
Immunogenicity | 10 months
  * Proportion of participants with VRC01-class IgG B-cells
  * Frequency of VRC01-class B-cells among IgG B-cells in PBMCs or in germinal centers, after each IP administration and at baseline
  * Proportion of participants with serum binding antibody responses to eOD-GT8 60mer, eOD-GT8 monomer, Core-g28v2 60mer, Core-g28v2 monomer, the CD4bs epitope on eOD-GT8, and the CD4bs epitope on Core-g28v2 after each IP administration and at baseline
  * Magnitude of responses to eOD-GT8 60mer, eOD-GT8 monomer, Core-g28v2 60mer, Core-g28v2 monomer, the CD4bs epitope on eOD-GT8, and the CD4bs epitope on Core-g28v2 after each IP administration and at baseline

OTHER OUTCOMES:
Exploratory Immunogenicity | 10 months
  * Analysis of overall mutation levels in VRC01 class IgG BCRs after each IP administration and at baseline, to assess overall maturation
  * Analysis of mutations in VRC01 class IgG BCRs to determine if they are conducive for development of VRC01-class bnAbs
  * Binding affinity and specificity of VRC01-class and non-VRC01-class vaccine induced antibodies identified by B-cell sorting and BCR sequencing after each IP administration, for eOD-GT8 and Core g28v2, and for candidate boost immunogens
  * Proportion of participants with serum antibody binding responses to Lumazine synthase, and magnitude of such responses, after each IP administration and at baseline
  * Proportion of participants with CD4 T-cell responses to eOD-GT8, Core-g28v2, and Lumazine synthase after each IP administration, and magnitude and epitope mapping of such responses
  * Proportion of participants with neutralization antibodies against tier 1 or 2 viral strains
  * Genotype of antibody gene alleles
  * Additional exploratory

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - UT Health San Antonio, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
To be Determined